CLINICAL TRIAL: NCT02107183
Title: Impact of Nasal High-flow vs Venturi Mask Oxygen Therapy on Weaning Outcome: a Multicenter, Randomized, Controlled Trial
Acronym: RINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Salvatore Maurizio MAGGIORE, MD, PhD, Associate Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Trial120_A
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Weaning Failure; Acute Respiratory Failure
Keywords: Oxygen therapy; Extubation; Weaning; Reintubation; Acute respiratory failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal high-flow oxygen therapy (Experimental): High-flow, fully humidified oxygen delivered through nasal cannula (Optiflow, Fisher & Paykel Healthcare) after extubation up to ICU discharge
  Interventions: Device: Optiflow (Fisher & Paykel Healthcare)
- Venturi mask oxygen therapy (Active Comparator): Oxygen delivered through standard Venturi mask after extubation up to ICU discharge
  Interventions: Device: Venturi mask

INTERVENTIONS:
Device: Optiflow (Fisher & Paykel Healthcare) — This device delivers high-flow oxygen through nasal cannula
  Arms: Nasal high-flow oxygen therapy
Device: Venturi mask — This device delivers low-flow oxygen at predetermined concentrations
  Arms: Venturi mask oxygen therapy

SUMMARY:
The purpose of this study is to determine whether, as compared with the Venturi mask, a nasal, high-flow oxygenation device (Optiflow) may reduce the extubation failure rate in patients needing oxygen therapy after extubation.

DETAILED DESCRIPTION:
This study compares the effects of two devices for oxygen therapy, the nasal, high-flow (Optiflow, intervention) and the Venturi mask (control), on the outcome of extubation. Available data suggest that Optiflow can improve oxygenation and patient's comfort in critically ill patients after extubation. The study hypothesis is that Optiflow may reduce the extubation failure rate in these patients.

In the intervention group, patients fulfilling inclusion criteria and not presenting any of the exclusion criteria will receive high-flow oxygen through nasal cannula (Optiflow, Fisher & Paykel Healthcare Ltd., New Zealand) after extubation. The oxygen concentration (FiO2) will be set to reach an oxygenation target similar to control patients (see below), while the gas flow rate will be set at 50 L/min.

In the control group, patients fulfilling inclusion criteria and not presenting any of the exclusion criteria will receive oxygen through a standard Venturi mask after extubation. The FiO2 will be set to obtain a arterial oxygen saturation (SpO2) between 92% and 98% (or between 88% and 95% in hypercapnic patients). Further FiO2 modifications will be performed by the attending physicians to meet the oxygenation target.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Mechanical ventilation > 24 hours
3. Signed Informed Consent
4. Successful spontaneous breathing trial
5. PaO2/FiO2 ratio ≤ 300 (or SpO2/FiO2 ratio ≤ 300 if SpO2 is lower than 98%) within 30 min after extubation while breathing through a Venturi mask with a delivered FiO2 of 31%

Exclusion Criteria:

1. Pregnancy
2. Presence of tracheostomy
3. Need for immediate post-extubation Non-Invasive Ventilation (>3 consecutive failures of the spontaneous breathing trial and/or a PaCO2 > 45 mmHg before the spontaneous breathing trial, with a respiratory rate ≥ 25/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reintubation | within 72 hours after extubation or at ICU discharge

SECONDARY OUTCOMES:
Need for Non-Invasive Ventilation | at day 28 after inclusion in the study or at ICU discharge
ICU length of stay | at day 28 from the inclusion in the study or at ICU discharge
Hospital length of stay | at day 28 from the inclusion in the study or at hospital discharge
ICU readmission | at day 28 from inclusion in the study
ICU mortality | at day 28 from inclusion in the study
Hospital mortality | at day 28 from inclusion in the study

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Maurizio Maggiore, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart, A. Gemelli Hospital, Rome, Italy
Locations (14):
- France (7):
  - Sainte-Marguerite University Hospital, Marseille
  - Lapeyronie University Hospital, Montpellier
  - Saint Eloi University Hospital, Montpellier
  - La Pitie-Salpetriere University Hospital, Paris
  - Louis Mourier University Hospital, Paris
  - Saint-Louis University Hospital, Paris
  - University Hospital, Poitiers
- Evangelismos University Hospital, Athens, Greece
- Italy (5):
  - Policlinico University Hospital, Bari
  - Università del Piemonte Orientale, Ospedale della Carità, Novara
  - Catholic University of the Sacred Heart, A. Gemelli Hospital, Rome
  - Le Molinette University Hospital, Turin
  - Università del Piemonte Orientale, Sant'Andrea Hospital, Vercelli
- Sant Pau University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Derived] Grieco DL, Jaber S, Zakynthinos S, Demoule A, Ricard JD, Navalesi P, Vaschetto R, Hraiech S, Klouche K, Frat JP, Lemiale V, Fanelli V, Chanques G, Longhini F, Mancebo J, Gualano MR, Ferreyro BL, Brochard LJ, Antonelli M, Maggiore SM; RINO trial study group. Use of rescue noninvasive ventilation for post-extubation respiratory failure. Crit Care. 2025 Nov 4;29(1):470. doi: 10.1186/s13054-025-05689-w. PMID 41188988
- [Derived] Maggiore SM, Jaber S, Grieco DL, Mancebo J, Zakynthinos S, Demoule A, Ricard JD, Navalesi P, Vaschetto R, Hraiech S, Klouche K, Frat JP, Lemiale V, Fanelli V, Chanques G, Natalini D, Ischaki E, Reuter D, Moran I, La Combe B, Longhini F, De Gaetano A, Ranieri VM, Brochard LJ, Antonelli M; RINO Trial Study Group. High-Flow Versus VenturiMask Oxygen Therapy to Prevent Reintubation in Hypoxemic Patients after Extubation: A Multicenter Randomized Clinical Trial. Am J Respir Crit Care Med. 2022 Dec 15;206(12):1452-1462. doi: 10.1164/rccm.202201-0065OC. PMID 35849787
- [Derived] Chaudhuri D, Granton D, Wang DX, Einav S, Helviz Y, Mauri T, Ricard JD, Mancebo J, Frat JP, Jog S, Hernandez G, Maggiore SM, Hodgson C, Jaber S, Brochard L, Burns KEA, Rochwerg B. Moderate Certainty Evidence Suggests the Use of High-Flow Nasal Cannula Does Not Decrease Hypoxia When Compared With Conventional Oxygen Therapy in the Peri-Intubation Period: Results of a Systematic Review and Meta-Analysis. Crit Care Med. 2020 Apr;48(4):571-578. doi: 10.1097/CCM.0000000000004217. PMID 32205604